CLINICAL TRIAL: NCT04661930
Title: A Study of a 10-days Fenofibrate Treatment, or Until Discharge From Hospital, Among COVID-19 Infected Patients Requiring Hospitalization
Brief Title: Fenofibrate for Patients With COVID-19 Requiring Hospitalization
Acronym: FENOC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yaakov Nahmias (Other)
Collaborators: Barzilai Medical Center (Other); Rambam Health Care Campus (Other); Nazareth Hospital (Other)
Responsible Party: Sponsor-Investigator, Yaakov Nahmias, Director of the Grass Center for Bioengineering, Hebrew University of Jerusalem
Organization: Hebrew University of Jerusalem (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0105-20-BRZ; FENOC-005
Record Dates: First submitted 2020-12-09; First posted 2020-12-10 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Corona Virus Disease (COVID-19); Respiratory Distress Syndrome; SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome | interventions — Fenofibrate

STUDY DESIGN:
Intervention Model Description: An interventional single-arm non-randomized pilot study in 15 patients, followed by an Interventional double-blinded randomized quadruple masked study in 40 patients.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Fenofibrate + Usual Care (Experimental): Participants in this arm will receive the study drug, Fenofibrate, in combination with usual care.
  Interventions: Drug: TriCor® 145mg tablets; Other: Usual care
- Placebo + Usual Care (Placebo Comparator): Participants in this arm will receive placebo treatment, in combination with usual care.
  Interventions: Other: Placebo; Other: Usual care
- Usual Care (Observetional) (No Intervention): Participants in this arm will receive the usual care and be compared by their medical records and laboratory results

INTERVENTIONS:
Drug: TriCor® 145mg tablets — Fenofibrate; 145 mg daily (1/day); oral administration; 10 days
  Other Names: Lipanthyl NT 145mg tablets
  Arms: Fenofibrate + Usual Care
Other: Placebo — Placebo (microcrystalline methylcellulose, gelatin capsule); oral administration
  Arms: Placebo + Usual Care
Other: Usual care — All participants will otherwise receive usual medical care
  Arms: Fenofibrate + Usual Care; Placebo + Usual Care

SUMMARY:
This is an open-label run-in followed by a randomized, double-blind drug treatment study of COVID-19 infected patients requiring inpatient hospital admission.

DETAILED DESCRIPTION:
This is an open-label run-in followed by a randomized, double-blind drug treatment study of COVID-19 infected patients requiring inpatient hospital admission. Open-label patients will be matched at least 1:10 with observational retrospective Propensity score-matched (PSM) patients' medical files. The double-blinded step will be randomized 2:1 to daily Fenofibrate or placebo for 10 days or hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Presumptive positive laboratory test for SARS-CoV-2 based on local laboratory standard
* Age greater than or equal to 18 years of age
* Severe COVID-19, defined by:

  * A disease severity score of 3 (Hospitalized, on non-invasive ventilation or high flow oxygen devices) to 4 (Hospitalized, requiring supplemental oxygen).

AND o A respiratory SOFA >=1 and increased oxygen requirement compared to baseline among those on home O2, a blood oxygen saturation of 93% or less on room air, a ratio of the partial pressure of oxygen to the fraction of inspired oxygen (PaO2/FiO2) of less than 300 mm Hg, respiratory rate >30 breaths/min, or lung infiltrates >50% on chest CT

• Enrollment within 72 hours of presentation of hospital admission or within 72 hours of a positive test result, whichever is later

Exclusion Criteria:

* Enrollment > 72 hours of admission order or positive test result, whichever is later
* Admission to the hospital with a respiratory SOFA >=5 , Critical COVID-19, or Disease Severity Score >5 (requiring extracorporeal membrane oxygenation (ECMO), invasive mechanical ventilation, or all)
* Known hypersensitivity to fenofibrate
* For female subjects:

  1. Pregenant, determined by a human chorionic gonadotropin (HCG) rapid detection kit or a blood test
  2. Breastfeeding
  3. Undergoing fertility treatments
* Patient-reported history or electronic medical record history of kidney disease, defined as:

  1. Any history of dialysis
  2. History of chronic kidney disease stage IV
  3. Estimated Glomerular Filtration Rate (eGFR) of < 30ml/min/1.73 m2 at the time of enrollment
* Acute pre-renal azotemia at the time of enrollment in the opinion of the investigator or bedside clinician
* Most recent mean arterial blood pressure prior to enrollment <65 mmHg
* Patient-reported history or electronic medical record history of severe liver disease, defined as:

  1. Cirrhosis
  2. History of hepatitis B or C
  3. Documented AST or ALT > 10 times the upper limit of normal measured within 24 hours prior to enrollment
* Patient-reported history or electronic medical record history of gallbladder disease
* Potassium >5.0 within 24 hours prior to enrollment unless a repeat value was <=5.0
* Treatment with coumarin anticoagulants (e.g., Warfarin), immunosuppressants (e.g. cisplatin), bile acid resins, or sulfonylurea.
* Inability to obtain informed consent from participant or legally authorized representative
* Enrollment in another blinded randomized clinical trial for COVID

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of Therapeutic Oxygen-Free Days | 14 days
  Outcome reported as the mean number of days participants in each arm did not require therapeutic oxygen usage during an in-patient hospital admission.
Length of Hospital Stay | 14 days
  Outcome reported as the mean length of in-patient hospital stay (in days) for participants in each arm
Viral Clearance by Nasopharyngeal Swab | 14 days
  Nasopharyngeal swabs will be collected every second day for the duration of study participation. Viral clearance is measured as fold change in viral genetic copies per mL
Difference in Estimated P/F Ratio at 14 days | 14 days
  Outcome calculated from the partial pressure of oxygen or peripheral saturation of oxygen by pulse oximetry divided by the fraction of inspired oxygen (PaO2 or SaO2 : FiO2 ratio). PaO2 is preferentially used if available.
Difference in Plasma Neutrophils at 14 days | 14 days
  Blood will be collected every second day for the duration of study participation. Difference will be calculated based on the first measurement after admission to the study.
Difference in Plasma Lymphocytes at 14 days | 14 days
  Blood will be collected every second day for the duration of study participation. Difference will be calculated based on the first measurement after admission to the study.
Difference in Plasma Monocytes at 14 days | 14 days
  Blood will be collected every second day for the duration of study participation. Difference will be calculated based on the first measurement after admission to the study.
Difference in Plasma C-Reactive Protein (CRP) at 14 days | 14 days
  Blood will be collected every second day for the duration of study participation. Difference will be calculated based on the first measurement after admission to the study.
Difference in Plasma IL-6 at 14 days | 14 days
  Blood will be collected every second day for the duration of study participation. Difference will be calculated based on the first measurement after admission to the study.
Difference in Plasma Procalcitonin (PCT) at 14 days | 14 days
  Blood will be collected every second day for the duration of study participation. Difference will be calculated based on the first measurement after admission to the study.
Difference in Plasma Ferritin at 14 days | 14 days
  Blood will be collected every second day for the duration of study participation. Difference will be calculated based on the first measurement after admission to the study.
Difference in NLR (Neutrophils to Lymphocytes Ratio) at 14 days | 14 days
  Blood will be collected every second day for the duration of study participation. Difference will be calculated based on the first measurement after admission to the study.

SECONDARY OUTCOMES:
14-Day Mortality | 14 days
  Outcome reported as the number of participants who have expired at 14 days post enrollment.
Difference in Organ Injury Plasma markers at 14 days - Lactate | 14 days
  Blood will be collected every second day for the duration of study participation. Difference will be calculated based on the first measurement after admission to the study.
Difference in Organ Injury Plasma markers at 14 days - Cardiac Troponin (TRO) | 14 days
  Blood will be collected every second day for the duration of study participation. Difference will be calculated based on the first measurement after admission to the study.
Difference in Organ Injury Plasma markers at 14 days - Creatine Kinase (CK) | 14 days
  Blood will be collected every second day for the duration of study participation. Difference will be calculated based on the first measurement after admission to the study.
Difference in Organ Injury Plasma markers at 14 days - Alanine Aminotransferase (ALT) | 14 days
  Blood will be collected every second day for the duration of study participation. Difference will be calculated based on the first measurement after admission to the study.
Difference in Organ Injury Plasma markers at 14 days - Alkaline Phosphatase (ALP) | 14 days
  Blood will be collected every second day for the duration of study participation. Difference will be calculated based on the first measurement after admission to the study.
Difference in Organ Injury Plasma markers at 14 days - D-dimer | 14 days
  Blood will be collected every second day for the duration of study participation. Difference will be calculated based on the first measurement after admission to the study.
Difference in Organ Injury Plasma markers at 14 days - Platelets (PLT) | 14 days
  Blood will be collected every second day for the duration of study participation. Difference will be calculated based on the first measurement after admission to the study.
Number of Abnormal Biomarker Days - D-dimer | 14 days
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Number of Abnormal Biomarker Days - Neutrophils | 14 days
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Number of Abnormal Biomarker Days - Lymphocytes | 14 days
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Number of Abnormal Biomarker Days - Platelets (PLT) | 14 days
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Number of Abnormal Biomarker Days - Monocytes | 14 days
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Number of Abnormal Biomarker Days - C-Reactive Protein (CRP) | 14 days
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Number of Abnormal Biomarker Days - IL-6 | 14 days
  Outcome reported as the mean number of days participants in each arm had 2 or more abnormal plasma levels.
Number of Abnormal Biomarker Days - Procalcitonin (PCT) | 14 days
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Number of Abnormal Biomarker Days - Lactate | 14 days
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Number of Abnormal Biomarker Days - Cardiac Troponin (TRO) | 14 days
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Number of Abnormal Biomarker Days - Creatine Kinase (CK) | 14 days
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Number of Abnormal Biomarker Days - Alanine Aminotransferase (ALT) | 14 days
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Number of Abnormal Biomarker Days - Alkaline Phosphatase (ALP) | 14 days
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Number of Abnormal Biomarker Days - Ferritin | 14 days
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Difference in Oxygenation at 14 days | 14 days
  PaO2 or SaO2 and FiO2. Partial pressure of oxygen or peripheral saturation of oxygen by pulse oximetry. FiO₂ is estimated from oxygen flow/delivery rates
Difference in Estimated PEEP adjusted P/F Ratio at 14 days | 14 days
  Outcome calculated from the partial pressure of oxygen or peripheral saturation of oxygen by pulse oximetry divided by the fraction of inspired oxygen (PaO2 or SaO2 : FiO2 ratio) and Expiratory Pressure.
Daily Hypotensive Episodes | 14 days
  Outcome reported as the mean number of daily hypotensive episodes (MAP < 65 mmHg) prompting intervention (indicated by a fluid bolus >=500 mL, new treatment with pressures, increase in 50% pressure or fluid rate) per participant in each arm.
Hypotension Requiring Vasopressors | 14 days
  Outcome reported as the number of participants in each arm requiring the use of vasopressors for hypotension.
Acute Kidney Injury | 14 days
  Outcome reported as the number of participants in each arm who experience acute kidney injury as defined by the Kidney Disease Improving Global Outcomes (KDIGO) guidelines: Increase in serum creatinine by 0.3mg/dL or more within 48 hours OR Increase in serum creatinine to 1.5 times baseline or more within the last 7 days OR Urine output less than 0.5 mL/kg/h for 6 hours.
Sequential Organ Failure Assessment (SOFA) Total Score | 14 days
  The SOFA assessment is used to track a person's risk status during stay in the Intensive Care Unit (ICU). The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal, and neurological systems. Each organ system is assigned a point value from 0 (normal) to 4 (high degree of dysfunction/failure). Total score is calculated by entering patient data into a SOFA calculator, a widely available software. Total scores range from 0-24, with higher scores indicating greater risk of mortality.
Oxygen Saturation / Fractional Inhaled Oxygen (F/S) | 14 days
  Oxygen saturation (percent) is measured by pulse oximeter. Fraction of inspired oxygen (FiO2) (unitless) is the volumetric fraction of oxygen to other gases in respiratory support. The F/S ratio is unitless.
28-Day Mortality | 28 days
  Outcome reported as the number of participants who have expired at 28 days post enrollment.
90-Day Mortality | 90 days
  Outcome reported as the number of participants who have expired at 90 days post enrollment.
ICU Admission | 14 days
  Outcome reported as the number of participants in each arm who require admission to the Intensive Care Unit (ICU).
Number of Ventilator-Free Days | 14 days
  Outcome reported as the mean number of days participants in each arm did not require mechanical ventilation during an in-patient hospital admission.
Number of Vasopressor-Free Days | 14 days
  Outcome reported as the mean number of days participants in each arm did not require vasopressor usage during an in-patient hospital admission.
Length of ICU Stay | 14 days
  Outcome reported as the mean length of stay (in days) in the Intensive Care Unit (ICU) for participants in each arm.
Incidence of Respiratory Failure | 14 days
  Outcome reported as the number of participants requiring BiPAP OR high flow nasal cannula OR mechanical ventilation OR extracorporeal membranous oxygenation (ECMO) utilization during in-patient hospital care in each arm.
Change in PROMIS Dyspnea Functional Limitations | 14 days
  The PROMIS Dyspnea (shortness of breath) item banks and pools assess self-reported Functional Limitations, Severity, Activity Motivation, Activity Requirements, Airborne Exposure, Assistant Devices Resources, Characteristics, Emotional Response, Task Avoidance and Time Extension as they related to dyspnea. In the 33-item Functional Limitations bank, 33 daily activities are rated in terms of degree of difficulty while engaging in the activity over the past 7 days (0 = no difficulty, 1 = a little difficulty, 2 = some difficulty, 3 = much difficulty). Total scores range from 0 to 99, with higher scores reflecting greater functional limitations.
Change in PROMIS Dyspnea Severity | 14 days
  The PROMIS Dyspnea (shortness of breath) item banks and pools assess self-reported Functional Limitations, Severity, Activity Motivation, Activity Requirements, Airborne Exposure, Assistant Devices Resources, Characteristics, Emotional Response, Task Avoidance and Time Extension as they related to dyspnea. The 33-item Severity bank assesses the severity of difficulty breathing during various specific activities (the same 33 activities assessed in Dyspnea Functional Limitations). Each activity is rated in terms of degree of dyspnea (0 = no shortness of breath, 1 = mildly short of breath, 2 = moderately short of breath, 3 = severely short of breath) while engaging in the activity over the past 7 days. Total scores range from 0 to 99 with higher scores reflecting greater levels of dyspnea during daily activity.
Disease Severity Rating | 14 days
  Outcome reported as the number of participants in each arm who fall into each of 7 categories. Lower scores indicate greater condition severity. The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen; 6) Not hospitalized, limitation on activities; 7) Not hospitalized, no limitations on activities.
Viral Load by Nasopharyngeal Swab | 14 days
  Nasopharyngeal swabs will be collected every fourth day for the duration of study participation. Viral load is measured as number of viral genetic copies per mL.
Viral Load by Blood | 14 days
  Blood will be collected every third day for viral load assessment for the duration of study participation. Viral load is measured as number of viral genetic copies per mL.
Viral Clearance by Blood | 14 days
  Blood will be collected every third day for viral load assessment for the duration of study participation. clearance is measured as fold change in viral genetic copies per mL.
Abnormal Biomarkers after recovery - D-dimer | 1 day
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Abnormal Biomarkers after recovery - Neutrophils | 1 day
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Abnormal Biomarkers after recovery - Lymphocytes | 1 day
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Abnormal Biomarkers after recovery - Platelets (PLT) | 1 day
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Abnormal Biomarkers after recovery - Monocytes | 1 day
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Abnormal Biomarkers after recovery - C-Reactive Protein (CRP) | 1 day
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Abnormal Biomarkers after recovery - IL-6 | 1 day
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Abnormal Biomarkers after recovery - Procalcitonin (PCT) | 1 day
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Abnormal Biomarkers after recovery - Lactate | 1 day
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Abnormal Biomarkers after recovery - Cardiac Troponin (TRO) | 1 day
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Abnormal Biomarkers after recovery - Creatine Kinase (CK) | 1 day
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Abnormal Biomarkers after recovery - Alanine Aminotransferase (ALT) | 1 day
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Abnormal Biomarkers after recovery - Alkaline Phosphatase (ALP) | 1 day
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Abnormal Biomarkers after recovery - Ferritin | 1 day
  Outcome reported as the mean number of days participants in each arm had abnormal plasma levels.
Abnormal Oxygenation after recovery | 1 day
  Outcome reported as the mean number of participants in each arm had abnormal PaO2 or SaO2 and FiO2 levels at the end of quarantine period. Partial pressure of oxygen or peripheral saturation of oxygen by pulse oximetry. FiO₂ is estimated from oxygen flow/delivery rates
PROMIS Dyspnea Functional Limitations after recovery | 1 day
  The PROMIS Dyspnea (shortness of breath) item banks and pools assess self-reported Functional Limitations, Severity, Activity Motivation, Activity Requirements, Airborne Exposure, Assistant Devices Resources, Characteristics, Emotional Response, Task Avoidance and Time Extension as they related to dyspnea. In the 33-item Functional Limitations bank, 33 daily activities are rated in terms of degree of difficulty while engaging in the activity over the past 7 days (0 = no difficulty, 1 = a little difficulty, 2 = some difficulty, 3 = much difficulty). Total scores range from 0 to 99, with higher scores reflecting greater functional limitations. Measured at the end of quarantine period.
PROMIS Dyspnea Severity after recovery | 1 day
  The PROMIS Dyspnea (shortness of breath) item banks and pools assess self-reported Functional Limitations, Severity, Activity Motivation, Activity Requirements, Airborne Exposure, Assistant Devices Resources, Characteristics, Emotional Response, Task Avoidance and Time Extension as they related to dyspnea. The 33-item Severity bank assesses the severity of difficulty breathing during various specific activities (the same 33 activities assessed in Dyspnea Functional Limitations). Each activity is rated in terms of degree of dyspnea (0 = no shortness of breath, 1 = mildly short of breath, 2 = moderately short of breath, 3 = severely short of breath) while engaging in the activity over the past 7 days. Total scores range from 0 to 99 with higher scores reflecting greater levels of dyspnea during daily activity. Measured at the end of quarantine period.

OTHER OUTCOMES:
Significant post-acute incident diagnoses after recovery at 28-days | 1 day
  Incident rate per 1000 at 28-days in hospitalized COVID-19 is ascertained from hospital admission until 28-days or end of follow-up.
Significant post-acute incident diagnoses after recovery at 90-days | 1 day
  Incident rate per 1000 at 90-days in hospitalized COVID-19 is ascertained from hospital admission until 90-days or end of follow-up.
Significant post-acute incident diagnoses after recovery at 6-months | 1 day
  Incident rate per 1000 at 6-months in hospitalized COVID-19 is ascertained from hospital admission until 6-months or end of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Mayaan, MD, Principal Investigator — Barzilai Medical Center; Mahram Nassar, MD, Study Director — Barzilai Medical Center; Yaakov Nahmias, PhD, Principal Investigator — Hebrew University of Jerusalem
Locations (3):
- Israel (3):
  - Barzilai Medical Center, Ashkelon
  - Rambam Health Care Campus, Haifa
  - Nazareth Hospital EMMS, Nazareth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bornstein SR, Dalan R, Hopkins D, Mingrone G, Boehm BO. Endocrine and metabolic link to coronavirus infection. Nat Rev Endocrinol. 2020 Jun;16(6):297-298. doi: 10.1038/s41574-020-0353-9. PMID 32242089
- [Background] Ehrlich, A., Uhl, S., Ioannidis, K., Hofree, M., tenOever, B., and Nahmias, Y. (2020). The SARS-CoV-2 Transcriptional Metabolic Signature in Lung Epithelium. SSRN Electronic Journal.
- [Background] McBride CE, Machamer CE. Palmitoylation of SARS-CoV S protein is necessary for partitioning into detergent-resistant membranes and cell-cell fusion but not interaction with M protein. Virology. 2010 Sep 15;405(1):139-48. doi: 10.1016/j.virol.2010.05.031. Epub 2010 Jul 1. PMID 20580052
- [Background] Wu Q, Zhou L, Sun X, Yan Z, Hu C, Wu J, Xu L, Li X, Liu H, Yin P, Li K, Zhao J, Li Y, Wang X, Li Y, Zhang Q, Xu G, Chen H. Altered Lipid Metabolism in Recovered SARS Patients Twelve Years after Infection. Sci Rep. 2017 Aug 22;7(1):9110. doi: 10.1038/s41598-017-09536-z. PMID 28831119
- [Background] Yan B, Chu H, Yang D, Sze KH, Lai PM, Yuan S, Shuai H, Wang Y, Kao RY, Chan JF, Yuen KY. Characterization of the Lipidomic Profile of Human Coronavirus-Infected Cells: Implications for Lipid Metabolism Remodeling upon Coronavirus Replication. Viruses. 2019 Jan 16;11(1):73. doi: 10.3390/v11010073. PMID 30654597
- [Background] Yang JK, Lin SS, Ji XJ, Guo LM. Binding of SARS coronavirus to its receptor damages islets and causes acute diabetes. Acta Diabetol. 2010 Sep;47(3):193-9. doi: 10.1007/s00592-009-0109-4. Epub 2009 Mar 31. PMID 19333547
- [Background] Yuan S, Chu H, Chan JF, Ye ZW, Wen L, Yan B, Lai PM, Tee KM, Huang J, Chen D, Li C, Zhao X, Yang D, Chiu MC, Yip C, Poon VK, Chan CC, Sze KH, Zhou J, Chan IH, Kok KH, To KK, Kao RY, Lau JY, Jin DY, Perlman S, Yuen KY. SREBP-dependent lipidomic reprogramming as a broad-spectrum antiviral target. Nat Commun. 2019 Jan 10;10(1):120. doi: 10.1038/s41467-018-08015-x. PMID 30631056
- [Background] Zhu L, She ZG, Cheng X, Qin JJ, Zhang XJ, Cai J, Lei F, Wang H, Xie J, Wang W, Li H, Zhang P, Song X, Chen X, Xiang M, Zhang C, Bai L, Xiang D, Chen MM, Liu Y, Yan Y, Liu M, Mao W, Zou J, Liu L, Chen G, Luo P, Xiao B, Zhang C, Zhang Z, Lu Z, Wang J, Lu H, Xia X, Wang D, Liao X, Peng G, Ye P, Yang J, Yuan Y, Huang X, Guo J, Zhang BH, Li H. Association of Blood Glucose Control and Outcomes in Patients with COVID-19 and Pre-existing Type 2 Diabetes. Cell Metab. 2020 Jun 2;31(6):1068-1077.e3. doi: 10.1016/j.cmet.2020.04.021. Epub 2020 May 1. PMID 32369736
- [Derived] Ehrlich A, Ioannidis K, Nasar M, Abu Alkian I, Daskal Y, Atari N, Kliker L, Rainy N, Hofree M, Shafran Tikva S, Houri I, Cicero A, Pavanello C, Sirtori CR, Cohen JB, Chirinos JA, Deutsch L, Cohen M, Gottlieb A, Bar-Chaim A, Shibolet O, Mandelboim M, Maayan SL, Nahmias Y. Efficacy and safety of metabolic interventions for the treatment of severe COVID-19: in vitro, observational, and non-randomized open-label interventional study. Elife. 2023 Jan 27;12:e79946. doi: 10.7554/eLife.79946. PMID 36705566